CLINICAL TRIAL: NCT01971983
Title: Effect of Two Osteopathic Techniques on Thickness of Paravertebral Muscles of the Lumbar Spine: Randomized Controlled Trial
Brief Title: Effect of Two Osteopathic Techniques on Thickness of Paravertebral Muscles of the Lumbar Spine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Fagundes Angellos, Physiotherapist, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Osteo-ufcspa
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2013-10

CONDITIONS: Low Back Pain
Keywords: Low back pain; Spinal manipulation; Osteopathy; Muscle energy technique; Muscle thickness
MeSH Terms: conditions — Low Back Pain | interventions — Tocopherols; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HVLA (Experimental): The subjects allocated to this group will receive a 'High-velocity, low-amplitude (HVLA) technique over the lumbar spine.
  Interventions: Other: High-velocity, low-amplitude (HVLA)
- ME (Experimental): Subjects allocated to this group will receive a muscle energy (ME) technique.
  Interventions: Other: Muscle energy (ME)
- Sham group (Sham Comparator): The individuals allocated to this group received an intervention of the "sham". The sample of this group will consist of subjects with history of dysfunctions of the lumbar spine.
  Interventions: Other: Sham

INTERVENTIONS:
Other: High-velocity, low-amplitude (HVLA) — With the subject lying on his/her side, the therapist will rotate the patient's trunk, flex his/her hip and knee of the upper leg. The therapist positions his caudad forearm over the hip, while the cephalad forearm lies over the patient's shoulder. The therapist's hands will be positioned over the lumbar spine's spinous process to be manipulated.
  Other Names: Thrust manipulation
  Arms: HVLA
Other: Muscle energy (ME) — This technique involves the active movement of the patient to activate a specific musculature in order to move a bony segment of a given joint in a specific direction in relation to the adjacent bone. This technique aims to restore the restricted movement of the joint in question.
  Other Names: Mitchell's technique
  Arms: ME
Other: Sham — Individuals in this group received a sham intervention type, in order to simulate an intervention.
  Arms: Sham group

SUMMARY:
The objective of this randomized controlled trial is to describe the effect of two osteopathic techniques - "high velocity, low amplitude" (HVLA) and muscle energy (ME) - on thickness, activation, strength, pressure pain threshold (PPT) of the paravertebral muscles at the lumbar spine, as well as the peak plantar pressures immediately and after a two-day follow-up.

The muscle thickness of the paravertebral muscles at the lumbar spine, namely internal oblique, external oblique and transversus abdominis can be altered after the application of 'high-velocity low-amplitude'(HVLA)and 'muscle energy' (ME)techniques immediately and after a two-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* At least one episode of low back pain over the last three months; confirmation of lumbar spine dysfunction by an experienced osteopath; age between 18 and 40 years; do not have performed physical stress activities over the last 24 hours; do not be physically active (physical activity for at least three times a week); fulfill the orientations to the follow-up assessment.

Exclusion Criteria:

* History of surgery, fracture or fixation on the lumbar spine and/or the pelvis; being pregnant; signs of radiculopathy; disc herniation at the lumbar spine; degenerative process at the lumbar spine; have received any kind of manipulative treatments over the past four weeks;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness | immediate
  We will evaluate the muscle thickness of four muscles that comprises the paravertebral musculature at the lumbar spine: internal oblique, external oblique, lumbar multifidus and transversus abdominis.
Muscle thickness | Two days
  We will evaluate the muscle thickness of four muscles that comprises the paravertebral musculature at the lumbar spine: internal oblique, external oblique, lumbar multifidus and transversus abdominis.

SECONDARY OUTCOMES:
Pressure pain threshold | Immediate
  subjects will be evaluated regarding their pressure pain threshold (PPT) on the spinous process of all of the lumbar vertebrae.
Pressure pain threshold | Two days
  subjects will be evaluated regarding their pressure pain threshold (PPT) on the spinous process of all of the lumbar vertebrae.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo F Angellos, Physiotherapis, Principal Investigator — The Federal University of Health Sciences of Porto Alegre
Locations (1):
- Laboratory of Physiotherapy - The Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil